CLINICAL TRIAL: NCT01479881
Title: A Phase I, 2-panel, Open-label, Randomized, Cross-over Trial in Healthy Subjects to Investigate the Effect of TMC435 at Steady-state on the Pharmacokinetics of the Immunosuppressants Cyclosporine and Tacrolimus
Brief Title: A Study in Healthy Participants Investigating the Effect of TMC435 on the Pharmacokinetics of Immunosuppressants Cyclosporine and Tacrolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100686; TMC435-TIDP16-C120 (Other: Tibotec Pharmaceuticals, Ireland); 2011-003021-96 (EudraCT Number)
Record Dates: First submitted 2011-10-20; First posted 2011-11-28 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; TMC435; TMC435-TiDP16-C120; TMC435-C120; HCV; Hepatitis C; Hep C; Healthy participants
MeSH Terms: conditions — Hepatitis C | interventions — Tacrolimus; Simeprevir; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): a single 100-mg dose of cyclosporine, and after a wash out period of at least 10 days, TMC435 150 mg once daily (q.d.) for 10 days on Days 1 to 10, coadministered with a single 100-mg dose of cyclosporine on Day 7.
  Interventions: Drug: cyclosporine; Drug: TMC435
- 002 (Experimental): TMC435 150 mg once daily (q.d.) for 10 days on Days 1 to 10, coadministered with a single 100-mg dose of cyclosporine on Day 7 and after a wash out period of at least 10 days, a single 100-mg dose of cyclosporine.
  Interventions: Drug: cyclosporine; Drug: TMC435
- 003 (Experimental): a single 2-mg dose of tacrolimus on Day 1. After a wash out period of at least 10 days, participants will receive TMC435 150 mg q.d. for 12 days on Days 1 to 12, coadministered with a single 2-mg dose of tacrolimus on Day 7.
  Interventions: Drug: tacrolimus; Drug: TMC435
- 004 (Experimental): TMC435 150 mg q.d. for 12 days on Days 1 to 12, coadministered with a single 2-mg dose of tacrolimus on Day 7. After a wash out period of at least 10 days, participants receive a single 2-mg dose of tacrolimus.
  Interventions: Drug: tacrolimus; Drug: TMC435

INTERVENTIONS:
Drug: tacrolimus — a single 2-mg dose of tacrolimus (on Day 1 in treatment C and on Day 7 in treatment D).
  Arms: 003; 004
Drug: TMC435 — TMC435, 150 mg daily for 12 days (Days 1 to 12 in treatment D).
  Arms: 003; 004
Drug: cyclosporine — A single 100-mg dose of cyclosporine (on Day 1 of treatment A and on Day 7 of treatment B).
  Arms: 001; 002
Drug: TMC435 — TMC435, 150 mg daily for 10 days (Day 1 - 10 in treatment B).
  Arms: 001; 002

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 (administered once a day) on the single-dose pharmacokinetics of the immunosuppressants cyclosporine and tacrolimus in healthy participants. Cyclosporine and tacrolimus are immunosuppressants used to prevent transplant rejection and may therefore potentially be coadministered with TMC435 in patients infected with hepatitis C virus that undergo liver transplantation. We will also explore the short-term safety and tolerability following coadministration of TMC435 at steady-state and (1) cyclosporine or (2) tacrolimus after single dosing in healthy participants. Steady-state is a term that means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is a protease inhibitor (PI) and is being investigated for treatment of chronic hepatitis C virus (HCV) infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). This is a Phase I, open-label (both participant and investigator know the name of the medication given at a certain moment) trial in 28 healthy participants to investigate the effect of TMC435 at steady-state on the single dose pharmacokinetics of the immunosuppressants cyclosporine and tacrolimus. The trial population will consist of a total of 28 healthy participants, equally divided over 2 panels. In Panel 1, each participant will receive 2 treatments: a single 100-mg dose of cyclosporine on Day 1 and TMC435 150 mg once daily for 10 days on Days 1 to 10, coadministered with a single 100-mg dose of cyclosporine on Day 7. In Panel 2, each participant will receive 2 treatments: a single 2-mg dose of tacrolimus on Day 1 and TMC435 150 mg each day for 12 days on Days 1 to 12, coadministered with a single 2-mg dose of tacrolimus on Day 7. Safety and tolerability will be assessed during the study period and during follow up. Blood and urine safety samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, Day1, Day 2 (only panel 1), Day 7(only panel 2), Day 8 (only panel 2) and at the follow-up visit about 5 to 7 days after last TMC435 intake.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal for at least 2 years, OR be surgically sterile, OR be not heterosexually active for the duration of the study or have a vasectomized partner OR if of childbearing potential and heterosexually active, be practicing a highly effective method of birth control before entry, and agree to continue to use the same method of contraception throughout the study and for at least 30 days after the last administration of study drug(s).

Exclusion Criteria:

* A positive Human Immunodeficiency Virus (HIV)-1 or HIV-2 test at screening;
* A positive Hepatitis A, B and C test at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in the steady-state plasma concentration (PK) of cyclosporine and tacrolimus following co-administration with TMC435. | Measured on Day1 till and including Day 7 for panel 1, and till and including Day 13 for panel 2. Reference is Day 1 for panel 1 and Day 7 for panel 2.
  Change in the steady-state plasma PK of cyclosporine and tacrolimus following co-administration with TMC435. PK characteristics of cyclosporine and tacrolimus are determined based on their respective plasma levels at one time point (Day 1 and Day 7 for respectively panel 1 and panel 2) and at 17 other time points. Standard PK parameters such as C0h, Cmin, Cmax, Tmax, AUC24h etc. will be determined.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability when combining TMC435 (150 mg, q.d.) with cyclosporine or tacrolimus. | Up to Day 50.
  to explore the short-term safety and tolerability following coadministration of TMC435 at steady-state and (1) 100-mg dose cyclosporine or (2) 2-mg dose tacrolimus after single dosing in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (1):
- Merksem, Belgium